CLINICAL TRIAL: NCT05205382
Title: Assessing the Effect of Nicotine Reduction on ENDS User's Addiction and Exposures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R01DA053587 (NIH)
Record Dates: First submitted 2021-12-15; First posted 2022-01-25 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Electronic Cigarette Use
Keywords: Nicotine reduction
MeSH Terms: conditions — Vaping | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electronic cigarette pods (SREC or NJOY) with 5% nicotine concentration (Experimental): Participants will complete a lab visit where they will use 5% nicotine electronic cigarette pods ad libitum for up to 60 minutes.
  Interventions: Other: 5% nicotine
- Electronic cigarette pods (NJOY) with 3% nicotine concentration (Experimental): Participants will complete a lab visit where they will use 3% nicotine electronic cigarette pods ad libitum for up to 60 minutes.
  Interventions: Other: 3% nicotine
- Electronic cigarette pods (SREC) with 0% nicotine concentration (Experimental): Participants will complete a lab visit where they will use 0% nicotine electronic cigarette pods ad libitum for up to 60 minutes.
  Interventions: Other: 0% nicotine

INTERVENTIONS:
Other: 5% nicotine — Effects of e-cigarette pods (JUUL/NJOY/SREC) with 5% nicotine concentration nicotine concentration
  Arms: Electronic cigarette pods (SREC or NJOY) with 5% nicotine concentration
Other: 3% nicotine — Effects of e-cigarette pods (JUUL/NJOY) with 3% nicotine concentration
  Arms: Electronic cigarette pods (NJOY) with 3% nicotine concentration
Other: 0% nicotine — Effects of e-cigarette pods (SREC) with 0% nicotine concentration
  Arms: Electronic cigarette pods (SREC) with 0% nicotine concentration

SUMMARY:
The rapid increase of electronic nicotine delivery systems (ENDS) use by young people in the US and their potential to harm health, cause addiction, and serve as a risk for cigarette smoking or dual-use is alarming. The epidemic of ENDS use among young people in the US has been associated with the rise in popularity of ENDS products that are very efficient in delivering high doses of nicotine to users. Therefore, the investigators propose to study the effects of nicotine reduction (NR) on young ENDS users as a potential regulatory strategy to reduce the addictiveness and use of ENDS. The proposed studies are directly responsive to research priories identified by the FDA and specified in this RFA under Addiction; studying the "Impact of changes in tobacco product characteristics (e.g. nicotine formulation) on dependence". This project aims to provide an overview of this project's rationale significance divided into 1) scientific rationale and regulatory implications; 2) the need to respond to the rising trend of ENDS use among young people in the US; 3) the importance of reducing the addictiveness of ENDS; 4) the strength of our clinical and analytical lab approach for regulatory purposes; and 5) the strengths and weaknesses in the rigor of prior research about NR for ENDS.

DETAILED DESCRIPTION:
The use of electronic nicotine delivery systems (ENDS or e-cigarettes) has reached epidemic levels among young people in the United States (US). ENDS emit toxic substances, including nicotine that irreversibly affects the developing brain and leads to dependence and increased risk of cigarette smoking initiation. Evidence indicates that young people using ENDS are likely to accelerate use and become nicotine dependent. Some of the most popular ENDS among youth (e.g. JUUL with 5% nicotine liquid) deliver in one cartridge a nicotine dose equal to an entire pack of cigarettes, and many users are unaware of this substantial exposure and the related risk of addiction. On the other hand, nicotine reduction (NR) has been considered by the US Food and Drug Administration (FDA) as an important strategy to limit the addictiveness and use of tobacco products.

Now that the FDA regulates ENDS under the "deeming rule", such a strategy can be considered for these emerging tobacco products. However, the investigators still lack evidence on the expected effects of a range of NR levels on ENDS users at different stages of use trajectory. Using clinical and analytical lab methods, the investigators plan to compare among 5% nicotine ENDS users the effect of partial (3%) or total (nicotine-free, 0%) NR on users' dependence, satisfaction, clinical (e.g. BP, oximetry, lung functions, symptoms), puffing behavior, and exposure to toxicants. The investigators will recruit current ENDS users (n=120; 21-35 yrs), for a 2X2 within subject crossover lab study. The nicotine conditions (5%, 3%) or (0%,5%) x 2 times (pre-post) are the within-subject factors.

Therefore, the study is divided into 2 parts, whereby the first part will be 2x2 comparing NJOY 5% and 3% to test the effects of partial nicotine reduction, and the second part will be using the NIDA Standardized Research Electronic Cigarette (SREC) for Clinical Research 5% and 0% (placebo), to test the effect of the total reduction using the same pods and juices from the same manufacturer.

The investigators hypothesize that NR will be associated with less satisfaction, withdrawal suppression, and intention to use and that such an effect will be more pronounced in total compared to partial NR and among high compared to low-dependency users. The proposed studies aim to answer 3 main regulatory questions: 1) is NR a promising regulatory option to reduce ENDS addictiveness and use; 2) what is the effect of partial vs. total NR on compensatory puffing and exposure to nicotine and respiratory toxicants, and 3) what is the effect of NR on ENDS users at different stages of their use. Combined, these studies will give direct and standardized evidence on the potential of NR regulations to limit the addictiveness and use of ENDS, and to help predict any potential side effects of NR on ENDS users' exposure to harmful toxicants.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy individuals (determined by physical examination).
* Age of 21-35 years.
* Is willing to provide informed consent.
* Is willing to attend the lab as required by the study protocol.
* Electronic cigarette users (defined as using electronic cigarette either daily or occasionally in the past 30 days)
* Have abstained from electronic cigarette use for 12 hours prior to each session

Exclusion Criteria:

* Report smoking cigarettes regularly (> 5 cigarettes/month in the past year).
* Report regular use of any other tobacco/nicotine product (e.g.,hookah, pipes, cigars) in the past year.
* Women who are breast-feeding or test positive for pregnancy (by urinalysis at screening).
* Individuals with self-reported history of chronic disease or current psychiatric conditions.
* Individuals with history of or active cardiovascular disease, low or high blood pressure, seizures, and regular use of prescription medications (other than vitamins or birth control).
* Individuals that report current THC (marijuana) smoking/vaping.
* Individuals that report the use of non-commercial (i.e., street) e-cigarette liquid or products
* Individuals that report current EVALI or COVID-19 related symptoms (i.e., cough, shortness of breath, chest pain, nausea, vomiting, abdominal pain, diarrhea, fever, chills, or weight loss)
* Individuals that have or have been exposed to COVID-19 in the last 14 days.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Plasma nicotine | During the 2 participant visits. Blood will be taken 2 times in each electronic cigarette use session: before and after an approximately 60 minutes ad lib use period
  Change in plasma nicotine level.

SECONDARY OUTCOMES:
Minnesota Nicotine Withdrawal Scale | During participants' 2 study visits. Questionnaire will be administered 2 times in each electronic cigarette use session: before and after an approximately 60 minutes ad lib use period
  This scale is used to assess the extent to which product use reduces tobacco abstinence. symptoms, and consists of 11 items scored 0 - 100. These items are presented as Visual Analog Scale with item (measure) centered above a horizontal line anchored on the left with not at all and on the right with extremely.
Tiffany-Drobes Questionnaire of Smoking Urges | During participants' 2 study visits. Questionnaire will be administered 2 times in each electronic cigarette use session: before and after an approximately 60 minutes ad lib use period
  This scale is used to assess the extent to which product use reduces tobacco abstinence symptoms, and consists of 10 items that are scored 0 - 7. Rated on a 7-point Likert scale ranging from 0 (strongly disagree) to 6 (strongly agree).
Carbon monoxide levels | During participants' 2 study visits. Carbon monoxide levels will be measured 2 times in each electronic cigarette use session: before and after an approximately 60 minutes ad lib use period
  Change in carbon monoxide levels (in parts per million).
Harm perception | During participants' 2 study visits. Questionnaire will be administered after each of the 2 electronic cigarette use sessions. Each session is approximately 60 minutes ad lib use period
  This scale will assess waterpipe harm perception and measure perceptions of waterpipe. relative risk compared to cigarettes. The scale will be scored on a 7-point scale ranging from 1 (not at all harmful), to 7 (extremely harmful).
Duke Sensory Questionnaire | During participants' 2 study visits. Questionnaire will be administered after each of the 2 electronic cigarette use sessions. Each session is approximately 60 minutes ad lib use period
  This scale will assess participants sensory experience of the inhaled product. The scale has nine items. All items will be scored on a 7-point Likert scale anchored at the extremes (1= not at all; 7=extremely).
The Cigarette/ENDS Evaluation Scale (WES) | During participants' 2 study visits. Questionnaire will be administered after each of the 2 electronic cigarette use sessions. Each session is approximately 60 minutes ad lib use period
  This scale assesses participants' perception of ENDS use. The scale has 11 items. All items will be scored on a 7-point Likert scale anchored at the extremes (1= not at all; 7=extremely).
Lung function tests (LFTs) | During participants' 2 study visits. Lung function tests will be measured 2 times in each electronic cigarette use session: before and after an approximately 60 minutes ad lib use period
  LFTs (i.e., lung volume testing, airway resistance, specific airway conductance) will be measured before and immediately after ENDS use. According to 2019 American Thoracic Society and European Respiratory Society recommendation simple spirometry (e.g., % predicted value pred (FVC), FEV1 % pred FEV1/FVC, % pred); forced expiratory flow (FEF) and peak expiratory flow rate or (PEFR) will be performed. Diffusing capacity for carbon monoxide (DLCO) will be determined using a rapidly resolving gas analyzer (RGA) and the single-breath technique. Note: This outcome is not involved in multiple assessments since all the values will appear on the spirometry at the same time.
Puff topography | During participants' 2 study visits. Puffing behavior is continuously measured during each electronic cigarette use session (an approximately 60 minutes ad lib use period)
  Measurement of puffing behavior.
Toxicant exposure (nicotine and aldehydes) | During the 2 participant visits. Toxicant exposure will be measured 2 times in each electronic cigarette use session: before and after an approximately 60 minutes ad lib use period
  This aim will help elucidate how compensatory puffing behavior in response to NR affects exposure to pulmonary toxicants. The investigators hypothesize that partial but not total NR will be associated with compensatory puffing behavior that will, in turn, lead to greater exposure to toxicants. The analytical assessments will be conducted at the AUB Aerosol Research Laboratory (ARL).The ARL is equipped with gas chromatographs with a flame ionization detector and a mass spectrometer (GC-FID, GC-MS), as well as and High-performance liquid chromatography Mass Spectrometry (HPLC-MS) for nicotine and aldehydes analysis. ARL optimized analytical methods have been used in several NIH-funded studies of ENDS nicotine and aldehydes emissions.

OTHER OUTCOMES:
Heart rate | During participants' 2 study visits. Heat rate will be measured from baseline continuously throughout each approximately 60 minutes session
  Change in heart rate, measured in beats per minute.
Blood pressure | During participants' 2 study visits. Blood pressure will be measured from baseline continuously throughout each approximately 60 minutes session
  Change in blood pressure, measured in mm/hg.

CONTACTS AND LOCATIONS:
Overall Officials: Wasim Maziak, PhD, MD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferdous T, Roy S, Chowdhury S, Jebai R, Maya L, DeCaprio AP, Bursac Z, Maziak W. Partial Nicotine Reduction and E-Cigarette Users' Puffing Behaviors Among Adults Aged 21 to 35 Years: A Randomized Crossover Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2422954. doi: 10.1001/jamanetworkopen.2024.22954. PMID 39058490

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT05205382/Prot_SAP_003.pdf
  • Informed Consent Form (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT05205382/ICF_002.pdf